CLINICAL TRIAL: NCT04212429
Title: The Clinical Safety of Topical Levofloxacin 1.5% vs Topical Moxifloxacin 0.5%
Brief Title: The Clinical Safety of Levofloxacin 1.5% vs Topical Moxifloxacin 0.5%
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Collaborators: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Wan Haslina Wan Abdul Halim, Consultant Ophthalmologist-Cornea And Anterior Segment, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FF-2019-320
Record Dates: First submitted 2019-12-10; First posted 2019-12-27 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2019-12

CONDITIONS: Endophthalmitis Postoperative
Keywords: Clinical Safety; Levofloxacin 1.5%; Moxifloxacin 0.5%

STUDY DESIGN:
Intervention Model Description: The qualified patients will be randomized on a 1:1 ratio into each treatment arm. Qualified eyes were further randomized into one of four subgroups, which specified the time between the last drop of study medication and the time of aqueous and vitreous humor sample collection (i.e., 1-, 2-, 4-, and 6-hour subgroups- about 32 patients per subgroup. Within each subgroups, there will be 16 of Levofloxacin group and 16 of Moxifloxacin group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Levofloxacin -1 hour group (Active Comparator): Levofloxacin hydrate, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 1-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection.
  Interventions: Drug: Levofloxacin Ophthalmic Product
- Levofloxacin-2 hour group (Active Comparator): Levofloxacin hydrate, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 2-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection.
  Interventions: Drug: Levofloxacin Ophthalmic Product
- Levofloxacin-4 hour group (Active Comparator): Levofloxacin hydrate, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 4-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection.
  Interventions: Drug: Levofloxacin Ophthalmic Product
- Levofloxacin-6 hour group (Active Comparator): Levofloxacin hydrate, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 6-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection.
  Interventions: Drug: Levofloxacin Ophthalmic Product
- Moxifloxacin-1 hour group (Active Comparator): Moxifloxacin hydrochloride, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 1-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection.
  Interventions: Drug: Moxifloxacin Ophthalmic Solution
- Moxifloxacin-2 hour group (Active Comparator): Moxifloxacin hydrochloride, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 2-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection.
  Interventions: Drug: Moxifloxacin Ophthalmic Solution
- Moxifloxacin-4 hour group (Active Comparator): Moxifloxacin hydrochloride, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 4-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection.
  Interventions: Drug: Moxifloxacin Ophthalmic Solution
- Moxifloxacin-6 hour group (Active Comparator): Moxifloxacin hydrochloride, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 8-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection.
  Interventions: Drug: Moxifloxacin Ophthalmic Solution

INTERVENTIONS:
Drug: Levofloxacin Ophthalmic Product — Levofloxacin hydrate, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily for 3 days pre-operatively and one drop on the day of operation.
  Other Names: Cravit 1.5%
  Arms: Levofloxacin -1 hour group; Levofloxacin-2 hour group; Levofloxacin-4 hour group; Levofloxacin-6 hour group
Drug: Moxifloxacin Ophthalmic Solution — Moxifloxacin hydrochloride, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily for 3 days pre-operatively and one drop on the day of operation.
  Other Names: Vigamox 0.5%
  Arms: Moxifloxacin-1 hour group; Moxifloxacin-2 hour group; Moxifloxacin-4 hour group; Moxifloxacin-6 hour group

SUMMARY:
Endophthalmitis is defined as intraocular inflammatory disorder affecting the vitreous cavity that can result from exogenous or endogenous spread of infecting organisms into the eye. Patients presents with reduced or blurred vision, red eye, pain, and lid swelling.

Endophthalmitis can progress into panophthalmitis, corneal infiltration and perforation, and finally phthisis bulbi. For exogenous endopthalmitis, the intraocular inflammation occurs due to a breach of the ocular compartment. The infectious agent indirectly introduced into the eye. This usually happens after intraocular surgery such as cataract surgery, vitrectomy, glaucoma filtration surgery, intravitreal injections, and other causes include penetrating ocular trauma or from adjacent periocular tissue. Several prophylactic measures have been taken to reduce the incidence of post-operative endopthalmitis postcataract surgery, this includes the use of pre-operative topical levofloxacin, intrameral cefuroxime, and providone iodine as ocular surface preparation.The proposed study is to evaluate clinical safety of Levofloxacin 1.5% and Moxifloxacin 0.5% on the anterior segment parameters.

DETAILED DESCRIPTION:
This is a prospective, double - blinded randomized clinical trial conducted in University Kebangsaan Malaysia Medical Centre (UKMMC) where there are two intervention arms. All patients from Ophthalmology Clinic in UKM Medical Centre from September 2019 till December 2021 will be involved in this study. Patients who fulfill the inclusion criteria will be included in this study. All eligible subjects will be asked to sign an informed consent.

The qualified patients will be randomized on a 1:1 ratio into each treatment arm. Qualified eyes were further randomized into one of four subgroups, which specified the time between the last drop of study medication and the time of aqueous and vitreous humor sample collection (i.e., 1-, 2-, 4-, and 6-hour subgroups- about 32 patients per subgroup-: 16 Levofloxacin, 16 Moxifloxacin.

Patient will undergo clinical assessment at the outpatient Ophthalmology Clinic at UKMMC. Initially, a non-contact assessment of the corneal surface will be done by the Keratograph 5. The parameters recorded are non-invasive tear break up time (NITBUT), tear film properties and redness analysis. The endothelial cell count will be analysed with a specular microscopy. Subsequently, patient will be assessed by a blinded ophthalmologist for clinical evaluation of corneal surface which includes tear break up time (TBUT), ocular surface abnormality and Rose-bengal staining. During the first visit, each patient will be educated on proper instillation of the eye drops to ensure the proper dose is administered. A prior observation of self- instillation of the eye drop by the study staff is required.

For 3 days prior to the day of the elective vitrectomy surgery, subjects will instill exactly one drop of study medication into their operative eye four times daily. On the day of surgery (visit 2, day 4), patients will receive their final drop of study medication administered by trained study personnel at the study site.

Post-vitrectomy, patients will be continued on the specified antibiotics for 4 hourly for 2 weeks. Then the antibiotic will taper down to 6 hourly (QID) daily for 1 week and antibiotics will be discontinued after that. Corneal safety will be assessed at 1 week and 4 weeks post operatively.

ELIGIBILITY:
Inclusion Criteria:

* All patients planned for vitrectomy for macula hole, ERM, RD surgery
* Age 18 and above
* Not on any topical medication

Exclusion Criteria:

* Patients with underlying ocular surface disease
* Fluoroquinolone allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of change in corneal surface in patients treated with topical levofloxacin 1.5% ophthalmic solution and topical moxifloxacin 0.5% ophthalmic solution | Day 3 of eyedrop instillation
  Evaluation of non-invasive tear break-up time (NITBUT), redness analysis, tear meniscus height and Tear Break-up Time (TBUT) of corneal surface from Baseline by using Oculus Keratograph-5 Machine at Day 3 of eyedrop instillation. Corneal surface signs (ie punctate epithelial erosions) is also measured by slit-lamp examination and graded using Oxford Scale Eye Grading.
Comparison of change in corneal surface in patients treated with topical levofloxacin 1.5% ophthalmic solution and topical moxifloxacin 0.5% ophthalmic solution. | 1-month post operation
  Evaluation of non-invasive tear break-up time (NITBUT), redness analysis, tear meniscus height and Tear Break-up Time (TBUT) of corneal surface from Baseline by using Oculus Keratograph-5 Machine at 1-month post operation. Corneal surface signs (ie punctate epithelial erosions) is also measured by slit-lamp examination and graded using Oxford Scale Eye Grading.
Comparison of Concentration of Endothelial cell count (cells/mm2) in patients treated with topical levofloxacin 1.5% ophthalmic solution and topical moxifloxacin 0.5% ophthalmic solution | Day 3 of eyedrop instillation
  Change in Concentration of Endothelial cell count (cells/mm2) from Baseline, measured at Day 3 of eyedrop instillation using a non-contact TOPCON Specular Microscopy model SP-1P.
Comparison of Concentration of Endothelial cell count (cells/mm2) in patients treated with topical levofloxacin 1.5% ophthalmic solution and topical moxifloxacin 0.5% ophthalmic solution | 1-month post-operation
  Change in Concentration of Endothelial cell count (cells/mm2) from Baseline, measured at 1-month post-operation using a non-contact TOPCON Specular Microscopy model SP-1P.
Comparison of Endothelial cell morphology in patients treated with topical levofloxacin 1.5% ophthalmic solution and topical moxifloxacin 0.5% ophthalmic solution | Day 3 of eyedrop instillation
  Change in Endothelial cell morphology from Baseline by assessing the Polymegathism (CV) which is the variation in individual cell areas, and Pleomorphism which is the increased in variability of cell shape, at Day 3 of eyedrop instillation using a non-contact TOPCON Specular Microscopy model SP-1P.
Comparison of Endothelial cell morphology in patients treated with topical levofloxacin 1.5% ophthalmic solution and topical moxifloxacin 0.5% ophthalmic solution | 1-month post-operation
  Change in Endothelial cell morphology from Baseline by assessing the Polymegathism (CV) which is the variation in individual cell areas, and Pleomorphism which is the increased in variability of cell shape, at 1-month post-operation using a non-contact TOPCON Specular Microscopy model SP-1P.

SECONDARY OUTCOMES:
Side effects | Post-operative period until study completion, an average of 2 years
  To report any untoward incidence of endophthalmitis during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Wan Haslina Wan Abdul Halim, M.D(UKM), Study Chair — National University of Malaysia
Locations (1):
- UKM Medical Centre, Cheras, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Jackson TL, Paraskevopoulos T, Georgalas I. Systematic review of 342 cases of endogenous bacterial endophthalmitis. Surv Ophthalmol. 2014 Nov-Dec;59(6):627-35. doi: 10.1016/j.survophthal.2014.06.002. Epub 2014 Jun 18. PMID 25113611
- [Background] Nishida T, Ishida K, Niwa Y, Kawakami H, Mochizuki K, Ohkusu K. An eleven-year retrospective study of endogenous bacterial endophthalmitis. J Ophthalmol. 2015;2015:261310. doi: 10.1155/2015/261310. Epub 2015 Jan 31. PMID 25802752
- [Background] Kernt M, Kampik A. Endophthalmitis: Pathogenesis, clinical presentation, management, and perspectives. Clin Ophthalmol. 2010 Mar 24;4:121-35. doi: 10.2147/opth.s6461. PMID 20390032
- [Background] Puustjarvi T, Terasvirta M, Nurmenniemi P, Lokkila J, Uusitalo H. Penetration of topically applied levofloxacin 0.5% and ofloxacin 0.3% into the vitreous of the non-inflamed human eye. Graefes Arch Clin Exp Ophthalmol. 2006 Dec;244(12):1633-7. doi: 10.1007/s00417-006-0360-0. PMID 16715252
- [Result] Hariprasad SM, Blinder KJ, Shah GK, Apte RS, Rosenblatt B, Holekamp NM, Thomas MA, Mieler WF, Chi J, Prince RA. Penetration pharmacokinetics of topically administered 0.5% moxifloxacin ophthalmic solution in human aqueous and vitreous. Arch Ophthalmol. 2005 Jan;123(1):39-44. doi: 10.1001/archopht.123.1.39. PMID 15642810
- [Result] Robertson SM, Curtis MA, Schlech BA, Rusinko A, Owen GR, Dembinska O, Liao J, Dahlin DC. Ocular pharmacokinetics of moxifloxacin after topical treatment of animals and humans. Surv Ophthalmol. 2005 Nov;50 Suppl 1:S32-45. doi: 10.1016/j.survophthal.2005.07.001. PMID 16257309
- [Result] Bucci FA Jr, Nguimfack IT, Fluet AT. Pharmacokinetics and aqueous humor penetration of levofloxacin 1.5% and moxifloxacin 0.5% in patients undergoing cataract surgery. Clin Ophthalmol. 2016 May 2;10:783-9. doi: 10.2147/OPTH.S91286. eCollection 2016. PMID 27194905
- [Result] Jackson MA, Schutze GE; COMMITTEE ON INFECTIOUS DISEASES. The Use of Systemic and Topical Fluoroquinolones. Pediatrics. 2016 Nov;138(5):e20162706. doi: 10.1542/peds.2016-2706. PMID 27940800
- [Result] Watanabe R, Nakazawa T, Yokokura S, Kubota A, Kubota H, Nishida K. Fluoroquinolone antibacterial eye drops: effects on normal human corneal epithelium, stroma, and endothelium. Clin Ophthalmol. 2010 Oct 21;4:1181-7. doi: 10.2147/OPTH.S13672. PMID 21060669
- [Result] Hanscom TA. Postoperative endophthalmitis. Clin Infect Dis. 2004 Feb 15;38(4):542-6. doi: 10.1086/381262. Epub 2004 Jan 26. PMID 14765348